CLINICAL TRIAL: NCT01746693
Title: Neurovascular Coupling in Subjects With Amblyopia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Gerhard Garhofer, Assoc. Prof. PD Dr., Medical University of Vienna
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: OPHT-291012
Record Dates: First submitted 2012-12-07; First posted 2012-12-11 (Estimated); Last update posted 2022-04-07 (Actual); Status verified 2022-04

CONDITIONS: Amblyopia ex Strabismus; Amblyopia ex Anisometropia
Keywords: retinal vessel diameter; retinal oxygen saturation; high resolution functional and anatomical imaging; inner retinal function; flicker response
MeSH Terms: interventions — Laser-Doppler Flowmetry

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- amblyopia ex anisometropia (Experimental): 20 male and female volunteers with amblyopia ex anisometropia
  Interventions: Device: Dynamic Vessel Analyzer; Other: Laser Doppler Velocimetry; Device: 7-Tesla MRI; Other: Pattern electroretinography; Other: Fourier domain optical coherence tomography
- amblyopia ex strabismus (Experimental): 20 male and female volunteers with amblyopia ex strabismus
  Interventions: Device: Dynamic Vessel Analyzer; Other: Laser Doppler Velocimetry; Device: 7-Tesla MRI; Other: Pattern electroretinography; Other: Fourier domain optical coherence tomography
- control subjects (Experimental): 20 healthy male and female control subjects
  Interventions: Device: Dynamic Vessel Analyzer; Other: Laser Doppler Velocimetry; Device: 7-Tesla MRI; Other: Pattern electroretinography; Other: Fourier domain optical coherence tomography

INTERVENTIONS:
Device: Dynamic Vessel Analyzer — retinal vessel diameter, retinal oxygen saturation
Other: Laser Doppler Velocimetry — retinal blood flow velocity, retinal blood flow
Device: 7-Tesla MRI — High resolution functional and anatomical imaging of the visual pathway
Other: Pattern electroretinography — inner retinal function
Other: Fourier domain optical coherence tomography — Blood flow in retina.

SUMMARY:
Amblyopia is a developmental condition that is characterized by reduced vision of the eye due to the presence of a sensory impediment during visual development, such as strabismus (ocular misalignment) or anisometropia (unequal refractive error), occurring early in life. Recent studies in humans and animals point towards a cortical locus for the processing deficit in amblyopia, revealing sensory deficits at the signal cell level. If changes in retinal neuronal function are also present, is unknown.

Like in the brain, blood flow in the retina is coupled to neuronal activity. This phenomenon has been measured by different study groups with non invasive techniques in the brain and retina. It has been shown in previous studies that stimulating the retina with diffuse luminant flickering light increases retinal vessel diameter and blood flow. However, it is unknown whether this is also the case in the retina of amblyopic eyes. Additionally, the introduction of blood oxygen level dependent (BOLD) fMRI also makes it possible to directly access the vascular response in the brain to visual stimuli.

Therefore, the aim of the present study is to investigate the effect of luminant flickering light on retinal vessel diameter and retinal blood flow in subjects with amblyopia. Also, oxygen saturation in retinal vessels will be assessed as well as pattern ERG for assessment of retinal function. Additionally, a high resolution image of the visual pathway will be taken with 7 Tesla MRI to investigate whether anatomical or functional alterations are present.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged between 18 and 55 years
* Non-smokers (for at least 6 months)
* Normal findings in the medical history and physical examination unless the investigator considers an abnormality to be clinically irrelevant
* Normal ophthalmic findings except amblyopia on one eye resulting from anisometropia or strabismus with a visual acuity of Snellen ≤ 0.3 with best correction on the amblyopic eye and Snellen 0.9 or better in the contralateral eye (for subjects with amblyopia)
* Normal ophthalmic findings with visual acuity of Snellen ≥ 1.0 in both eyes (for control subjects)

Exclusion Criteria:

* Symptoms of a clinically relevant illness in the 3 weeks before the first study day
* Presence or history of a severe medical condition as judged by the clinical investigator
* Regular use of medication, abuse of alcoholic beverages, participation in a clinical trial in the 3 weeks preceding the study (except oral contraceptives)
* Blood donation during the previous three weeks
* Pregnancy, planned pregnancy or lactating
* Any metallic, electric, electronic or magnetic device or object not removable except dental fillings
* Claustrophobia
* Epilepsia, history or family history of seizures

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-03 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-09-02 (Estimated)

PRIMARY OUTCOMES:
Retinal Vessel Diameter in Response to Flickering Light (DVA) | once on the study day

SECONDARY OUTCOMES:
Retinal (arterial and venous) oxygen saturation | once on the study day
Retinal blood velocity in response to flickering light | once on the study day
High resolution functional and anatomical imaging of the visual pathway | once on the study day
Inner Retinal Function | once on the study day

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Clinical Pharmacology, Medical University of Vienna, Vienna, Austria